CLINICAL TRIAL: NCT04395677
Title: A Multicenter, Open Label, Single Arm Phase 2 Study of AB-106 in the Treatment of Locally Advanced and Metastatic NSCLC
Brief Title: A Study of AB-106 in Subjects With Advanced NSCLC Harboring ROS1 Fusion Gene
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nuvation Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-106-C203
Record Dates: First submitted 2020-05-12; First posted 2020-05-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AB-106 （DS-6051b） (Experimental): Single-arm trial whereby all consented, enrolled, eligible patients receive AB-106
  Interventions: Drug: AB-106

INTERVENTIONS:
Drug: AB-106 — Stage 1: 400mg QD for 3 patients and 600mg QD for 3 patients
  Stage 2: 600mg QD
  Other Names: DS-6051b

SUMMARY:
The purpose of the study is to evaluate safety, pharmacokinetics and efficacy of AB-106 monotherapy in the treatment of advanced NSCLC.

DETAILED DESCRIPTION:
This is a Phase II, multicenter, single-arm, open label study of AB-106 in the Chinese patients with advanced NSCLC harboring ROS1 fusion gene.The study will be divided into two stages. First stage (Stage I) is to determine the clinical optimal dose of AB-106, which will be evaluated at two dose levels (400 mg QD and 600mg QD), and the safety, tolerability and pharmacokinetics of AB-106 will be evaluated at the same time; Second stage (Stage II) is to evaluate the efficacy and safety of AB-106 at the clinical optimal dose determined from Stage I. It is expected that 6 patients with advanced NSCLC harboring ROS1 fusion will be enrolled in the first stage. About 167 patients with ROS1 fusion will be enrolled in the second stage and divided into two treatment cohorts (Cohort A & Cohort B). It is planned to enroll about 106 ROS1-TKI treatment naïve patients in Cohort A and about 67 crizotinib pre-treated patients in Cohort B. AB-106 will be administered 600mg once daily in 21-day cycles. Patients will continue with the study treatment until progression of disease as determined by the investigator. The frequency of tumor assessments is once every 2 treatment cycles through Cycle 9, then every 3 treatment cycles through Cycle 27 and every 4 treatment cycles thereafter.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for enrollment into the study:

1. ≥ 18 years of age
2. Histologically or cytologically confirmed locally advanced or metastatic NSCLC
3. Positivity of ROS1 fusion is determined by the local qualified laboratories by using the FISH, RT-PCR or NGS assay, and the subject must provide archival tumor tissue sample for the confirmation by a sponsor-designated central laboratory
4. The subject is either TKI treatment naïve(Cohort A)， or has disease progression following the treatment of crizotinib （Cohort B）
5. The patient with brain metastases is either asymptomatic, or neurologically stable for at least 2 weeks prior to study entry
6. Prior therapies (including chemotherapies [less than 3 lines of regimen], radiotherapy [except for palliative], or surgery) should be completed at least 2 weeks prior to study entry. The palliative radiotherapy (≤10 times) should be completed within 48 hours prior to study entry. Any acute toxic effect must be resolved to CTCAE Grade ≤1 except for alopecia
7. At least one measurable target tumor lesion (as accessed by RECIST v1.1) that has not been irradiated
8. ECOG Performance Status: 0 or 1
9. Patient with a life expectancy ≥ 3 months based on the judgement of investigators

Adequate organ functions defined by the following criteria：

* Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤2.5 x ULN; or ≤5 x ULN， if there is liver metastases involvement；
* Total serum bilirubin ≤1.5 x ULN；
* Absolute neutrophil count（ANC） ≥1500/µL；
* Platelet count≥100,000/µL；
* Hemoglobin≥8.0 g/dL；
* Serum creatinine ≤2 x ULN. 11. Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of the pertinent aspect of the study 12. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures 13. Male and female patients of childbearing potential must agree to sue effective methods of contraception throughout the study and for 90 days after the last dose of study medication.

Exclusion Criteria:

Patient presenting with any of the following criteria will not be included in the study：

1. Current participation in other therapeutic investigational studies
2. Previous participation in the treatment or clinical trials of other ROS1-TKIs (except for crizotinib)
3. Previous participation in the treatment and clinical trials of ALK or NTRK fusion gene targeted therapies.
4. Spinal cord compression unless the patient demonstrates good pain control and stabilization or recovery of neurological function, carcinomatous meningitis or leptomeningeal disease
5. Patients with interstitial fibrosis or interstitial lung disease
6. Any one of the following currently or in the previous 3 months: myocardial infarction, severe/unstable angina, coronary/ peripheral artery bypass graft, congestive heart failure or cerebrovascular accident including transient ischemic attack
7. Ongoing cardiac dysrhythmias of NCI CTCAE (v5.0) Grade≥2, uncontrolled atrial fibrillation of any grade, or QTc interval>470 microsec
8. Pregnancy or breastfeeding
9. Current use of food or drugs that are known strong CYP3A inhibitors, including (but not limited to) atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin, voriconazole, grapefruit or grapefruit juice.
10. Current use of drugs that are known strong CYP3A4 inducers, including (but not limited to) carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, and St John's Wort
11. Current use of drugs that are known CYP3A4 substrates with narrow therapeutic indices, including (but not limited to) dihydroergotamine, ergotamine, pimozide, astemizole, cisapride, and terfenadine.
12. Current use of drugs that are known to induce QTc prolongation
13. Systematic treatment with anti-cancer therapy, including any Traditional Chinese Medicine (TCM)with anti-tumor effect indicated in the prescription information.
14. Evidence of active malignancy (other than current NSCLC, non-melanoma skin cancer, in situ cervical cancer, and presumed cured prostate cancer) within the last 3 years
15. Clinically active viral disease with positivity of serum HIV, HBV, HCV, RPR testing
16. Difficult to swallow which may significantly impact drug absorption
17. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation in the judgement of investigator and sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Best overall response (BOR) by IRC | 6 months
  Best overall response (BOR) based on independent radiology review by Independent Review Committee(IRC) according to RECIST 1.1

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 25 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Rate of ECG QT Interval prolongation patients in all patients | 25 months
  After the medicine, the number of patients with ECG QT Interval and the rate of patients with clinical significant
Maximum Plasma Concentration [Cmax] | Day 1 to Cycle1Day15
  The Cmax of Cycle1Day1 and Cycle1Day15 will be assessed, (each cycle is 21 days)
Area under the curve from time zero to τ (dose interval τ is 24 h in this study) [AUCτ] | Day 1 to Cycle1Day15
  The AUCτ of Cycle1Day1 and Cycle1Day15 will be assessed, (each cycle is 21 days)
Average plasma concentration at steady state over dosing interval [Cav] | Day 1 to Cycle1Day15
  The Cav of Cycle1Day1 and Cycle1Day15 will be assessed, (each cycle is 21 days)
Trough plasma concentration [Ctrough] | Day 1 to Cycle1Day15
  The Cthrough of Cycle1Day1 and Cycle1Day15 will be assessed, (each cycle is 21 days)
Time to reach maximum plasma concentration [Tmax] | Day 1 to Cycle1Day15
  The Tmax of Cycle1Day1 and Cycle1Day15 will be assessed, (each cycle is 21 days)
Duration of Response(DOR) | 25 months
  Duration of Response(DOR) based on independent radiology review by Independent Review Committee(IRC) and investigator according to RECIST 1.1
Time to Response(TTR) | 6 months
  Time to Response(TTR) based on independent radiology review by Independent Review Committee(IRC) and investigator according to RECIST 1.1
Time to Progress(TTP) | 25 months
  Time to Progress(TTP) based on independent radiology review by Independent Review Committee(IRC) and investigator according to RECIST 1.1
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
Progression free Survival(PFS) | 25 months
  Progression free Survival(PFS) based on independent radiology review by Independent Review Committee(IRC) and investigator according to RECIST 1.1
Intracranial best overall response (IBOR) | 25 months
  Intracranial Best overall response (BOR) based on independent radiology review by Independent Review Committee(IRC) and Investigator according to RANO for intracranial lesion
Duration of intracranial response (IDOR) | 25 months
  Duration of intracranial response (IDOR) based on independent radiology review by Independent Review Committee(IRC) and Investigator according to RANO for intracranial lesion
Overall Survival(OS) | 51 months
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Oncology, Study Director — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perol M, Li W, Pennell NA, Liu G, Ohe Y, De Braud F, Nagasaka M, Felip E, Xiong A, Zhang Y, Fan H, Wang X, Li S, Lai RK, Ran F, Zhang X, Chen W, Bazhenova L, Zhou C. Taletrectinib in ROS1+ Non-Small Cell Lung Cancer: TRUST. J Clin Oncol. 2025 Jun;43(16):1920-1929. doi: 10.1200/JCO-25-00275. Epub 2025 Apr 3. PMID 40179330
- [Derived] Li W, Xiong A, Yang N, Fan H, Yu Q, Zhao Y, Wang Y, Meng X, Wu J, Wang Z, Liu Y, Wang X, Qin X, Lu K, Zhuang W, Ren Y, Zhang X, Yan B, Lovly CM, Zhou C. Efficacy and Safety of Taletrectinib in Chinese Patients With ROS1+ Non-Small Cell Lung Cancer: The Phase II TRUST-I Study. J Clin Oncol. 2024 Aug 1;42(22):2660-2670. doi: 10.1200/JCO.24.00731. Epub 2024 Jun 1. PMID 38822758